CLINICAL TRIAL: NCT02316132
Title: Confocal Endomicroscopy for the Detection of Food Intolerances in Patients With IBS: Add on Control Group: Does Stress Cause Similar Mucosal Changes to Food Antigens?
Brief Title: Confocal Laser Endomicroscopy, IBS and Stress
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No appropriate participants
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Mark Ellrichmann, Senior Consultant, Unit of Experimental Endoscopy, University Hospital Schleswig-Holstein
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: IBS stress
Record Dates: First submitted 2014-12-05; First posted 2014-12-12 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress (Active Comparator): Injection of corticotropin releasing factor
  Interventions: Drug: Stress
- Control (Placebo Comparator): Injection of 0.9% saline 10 ml
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Stress — Corticotropin-Releasing Hormone
  Other Names: CRH
  Arms: Stress
Drug: Control — Saline 0.9%
  Other Names: Saline
  Arms: Control

SUMMARY:
After standard endomicroscopy with fluorescein to investigate for dysplasia in Barrett's esophagus the endoscope will be forwarded into the 2nd part of the duodenum. Fluorescein is needed for CLE but is not part of the investigation.

Initial CLE baseline images will be taken to assure intact mucosa and allow later detailed baseline counts of intraepithelial lymphocytes (IEL) and epithelial breaks in the duodenal mucosa.

Thereafter, either 10 ml NaCl 0.9% or 100µg CRF topped up to 10ml with NaCL 0.9% (according to randomisation) will be injected intravenously. Endoscopist and assistant staff will be blinded to the randomisation. Subsequently, the gut surface will be examined for at least 5 min with endomicroscopy for any change in IEL, epithelial breaks/gaps with extrusion of fluorescein into the gut lumen and widening of intervillous space.

Post procedure mucosal fluid will be aspirated for assessment of mast cell tryptase and eosin catatonic protein (ECP), and 8 duodenal biopsies will be taken for 1) electron microscopy to visualise mast cell degranulation and 2) paraffin embedding for subsequent staining for mast cell tryptase to identify mast cell activation and numbers.

The procedure will take around 15 minutes in addition to the routine investigation performed prior to the study. A study outline is presented in figure 1.

Samples taken are the same amount as done in the previous food associated study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* No abdominal symptoms such as bloating and abdominal pain
* Barrett's esophagus
* Independent indication for confocal laser endomicroscopy for evaluation of Barrett's dysplasia
* Written informed consent for participation in this study

Exclusion Criteria:

* Any known other gastrointestinal disease including infection such as helicobacter pylori, Morbus Whipple or others, celiac disease, or chronic inflammatory bowel disease
* Active or recent GI Bleeding
* Stricture in the upper gastrointestinal tract
* Impaired renal function (Creatinine >1.2 mg/dL)
* Pregnancy or breast feeding
* Inability to obtain informed consent
* Known allergy to Methylene blue or Fluorescein
* Participation in other clinical trials within the last 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
visible marked increase of leaks/gaps with extrusion of fluorescein into the gut lumen. | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Annette Fritscher-Ravens, MD, PhD, Principal Investigator — University Hospital Schleswig-Holstein; Mark Ellrichmann, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- Interdisciplinary Endoscopy, University hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany